CLINICAL TRIAL: NCT06762743
Title: A Randomized, Open-Label, Two-Formulation, Two-Period, Crossover Bioequivalence Study of Oral Brivaracetam Solution Administered As a Single Dose Under Fasting and High-fat Meal Conditions in Healthy Subjects
Brief Title: Bioequivalence Study of Two Brivaracetam Oral Solutions in Healthy Adults Under Fasting and High-Fat Meal Conditions
Acronym: BE
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 240605-BLXT-HBE
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy (treatment Refractory)
Keywords: crossover; bioequivalence; Brivaracetam Oral Solution
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Intervention Model Description: A two-period, two-sequence crossover design where participants are randomly assigned to receive either the test or reference formulation in a fasted or fed state, with a washout period of seven days between treatments.
Masking Description: This is an open-label study; all participants and investigators are aware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting group (Experimental): Participants in fasting group will first receive a single oral dose of the test formulation of Brivaracetam oral solution in the first period, followed by a washout period, and then a single oral dose of the reference formulation of Brivaracetam oral solution in the second period.
  Interventions: Drug: Brivaracetam Oral Solution (Test Formulation); Drug: Brivaracetam Oral Solution (Reference Formulation)
- High-fat meal group (Experimental): Participants will first receive a single oral dose of the reference formulation of Brivaracetam oral solution in the first period, followed by a washout period, and then a single oral dose of the test formulation of Brivaracetam in the second period.
  Interventions: Drug: Brivaracetam Oral Solution (Test Formulation); Drug: Brivaracetam Oral Solution (Reference Formulation)

INTERVENTIONS:
Drug: Brivaracetam Oral Solution (Test Formulation) — The drug is manufactured by Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. The formulation is provided as a 300 mL: 3 g solution, with a dosage of 10 mL (100 mg) per single oral dose. The drug will be administered to participants in the fasting group during the first phase of the study and to participants in the high-fat meal group during the second phase of the study.
Drug: Brivaracetam Oral Solution (Reference Formulation) — The drug is manufactured by UCB Pharma S.A. under the trade name Briviact®. The formulation is provided as a 300 mL: 3 g solution, with a dosage of 10 mL (100 mg) per single oral dose. The drug will be administered to participants in the fasting group during the first phase of the study and to participants in the high-fat meal group during the second phase of the study.
  Other Names: Briviact®

SUMMARY:
The goal of this clinical trial is to evaluate the bioequivalence of Brivaracetam oral solution under fasting and high-fat meal conditions in healthy adults. The study will compare a test formulation (produced by Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd., 300ml: 3g) to the reference formulation (Briviact®, UCB Pharma S.A., 300ml: 3g).

The main questions it aims to answer are:

1. Do the test and reference formulations of Brivaracetam oral solution exhibit similar pharmacokinetic behavior in the body?
2. What are the clinical safety outcomes for participants taking the test and reference formulations?

Participants will:

Be randomly assigned to two treatment sequences (T-R or R-T) in a 1:1 ratio. Receive either the test formulation or reference formulation of Brivaracetam oral solution (10ml), taken with 240mL of warm water, under either fasting or high-fat meal conditions.

Cross over to the alternate formulation after a 7-day washout period, completing a total of two treatment periods (2 weeks).

Undergo regular checkups and tests to monitor pharmacokinetics and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age and Gender: Healthy male and female participants aged 18-55 years (inclusive).
* Weight and BMI: Male participants must weigh ≥50 kg, and females ≥45 kg, with a body mass index (BMI) between 19 and 26. BMI is calculated as: BMI = weight (kg) / height (m²).
* Participants must fully understand the purpose, methods, content, and test drugs of this study before enrollment, be capable of good communication with investigators, adhere to study requirements, and voluntarily sign the informed consent form.
* Participants must commit to avoiding pregnancy and refraining from sperm/egg donation from the time of consent through 3 months after the last dose. Participants must agree to use effective contraception (non-pharmacological methods) during the trial. Female participants must have had no unprotected sexual activity within 14 days before the first dose.

Exclusion Criteria:

* History of allergies (e.g., angioedema, anaphylactic shock) or hypersensitivity (e.g., to pollen, two or more drugs/foods), or known allergy to briciclib or its excipients.
* Past or current illnesses that may affect drug absorption, distribution, metabolism, excretion, or the interpretation of safety data, or conditions reducing compliance, including but not limited to gastrointestinal, renal, hepatic, pulmonary, neurological, hematological, endocrine, oncological, immunological, psychiatric, or cardiovascular diseases, as judged by the investigator.
* Major surgery within 3 months prior to screening or planned surgery during the study period, including procedures affecting pharmacokinetics (e.g., gallbladder/biliary tract surgery).
* History of significant bleeding, active bleeding, thrombocytopenia, coagulation disorders, or family history of coagulopathy.
* Vaccination within 28 days prior to screening or planned vaccination during the study.
* History of substance abuse or dependence within the past 5 years or use of drugs such as morphine, methamphetamine, ketamine, cannabis, or ecstasy within 6 months before screening. Positive urine drug screen results are also exclusionary.
* Difficulty with venipuncture, intolerance to venous puncture, or history of needle or blood phobia.
* Lactose intolerance.
* Special dietary requirements that cannot align with standardized study diets.
* Participation in any clinical trial and drug administration within 3 months prior to screening.
* Blood donation or significant blood loss (≥400 mL) within 3 months prior to screening (excluding physiological blood loss in women) or intention to donate blood during the study.
* Regular smokers (≥5 cigarettes/day) or habitual betel nut chewers within 3 months prior to screening, or inability to abstain from tobacco products during the study.
* Frequent alcohol consumption (more than 14 units per week, where 1 unit = 360 mL beer, 45 mL spirits, or 150 mL wine) within 3 months prior to screening, positive breath alcohol test, or inability to abstain from alcohol during the study.
* Excessive intake of tea, coffee, caffeine-containing products, grapefruit, or xanthine-rich foods or beverages (e.g., theophylline, caffeine, theobromine) averaging more than 8 cups/day (1 cup = 200 mL) within 3 months prior to screening or inability to discontinue such intake during the study.
* Use of any medications, including prescription, over-the-counter drugs, herbal medicines, or health supplements, within 14 days prior to the first dose.
* Use of any liver enzyme-altering drugs within 28 days prior to the first dose.
* Pregnant or lactating women, or females with positive pregnancy tests.
* Positive results for any of the following virological tests: Hepatitis B surface antigen, Hepatitis C antibody, HIV antibody, or syphilis antibody.
* Clinically significant abnormalities in physical examination, vital signs, 12-lead ECG, or laboratory tests at screening, as determined by the investigator.
* Other reasons that may prevent the participant from completing the study, or any other factors deemed unsuitable for participation by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | two weeks
  Cmax is the maximum observed plasma concentration of the drug following a single oral dose. This parameter reflects the peak exposure to the drug in the bloodstream after administration.
Area Under the Plasma Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-t) | two weeks
  AUC0-t represents the total drug exposure from time 0 to the last measurable concentration. It is an important pharmacokinetic parameter for understanding the extent of drug absorption over time.
Area Under the Plasma Concentration-Time Curve from Time 0 to Infinity (AUC0-∞) | two weeks
  AUC0-∞ is the area under the plasma concentration-time curve from time 0 to infinity, capturing the total exposure to the drug. It includes all measurable concentrations, both during and after the absorption phase.

SECONDARY OUTCOMES:
Time to Reach Maximum Plasma Concentration(Tmax ) | two weeks
  Tmax is the time it takes to reach the maximum plasma concentration (Cmax) after a single dose of the drug. It indicates the rate at which the drug is absorbed into the bloodstream.
Terminal Elimination Rate Constant (λz) | two weeks
  λz is the terminal elimination rate constant, which is used to describe the rate at which the drug is cleared from the body during the elimination phase. This value helps estimate the half-life of the drug.
Half-life (t1/2) | two weeks
  t1/2 is the time required for the plasma concentration of the drug to decrease by half. It is a key pharmacokinetic parameter to understand the duration of action of the drug.
Percentage of the Area Under the Curve Extrapolated to Infinity(AUC_%Extrap ) | two weeks
  AUC_%Extrap is the percentage of the total AUC that is extrapolated beyond the last measured concentration (AUC∞ - AUC0-t) / AUC∞. This indicates the reliability of the AUC data and how much data is based on extrapolated values.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: IPD and supporting information will be available starting from the publication of the primary study results.
  End Date: IPD and supporting information will be available for a period of five years following the study's completion and publication. After this period, access may be restricted or subject to specific conditions.
Access Criteria: Qualified researchers, including academic institutions, non-profit organizations, and industry collaborators, will be able to access the de-identified individual participant data (IPD), provided they meet the necessary data use requirements.
  The available IPD will include the de-identified clinical and laboratory data collected throughout the study, such as demographic information, baseline clinical characteristics, treatment regimens, and efficacy and safety outcomes, including adverse events, pharmacokinetic data, and biomarker analyses.
  Data will be made available upon request through https://clinicalstudydatarequest.com/. Researchers wishing to access the data must submit a formal request, which will be evaluated based on the study's data sharing policies and relevant data use agreements.

REFERENCES:
- [Background] Velazquez J, Acosta J, Herrera N, Morales A, Gonzalez O, Herrera F, Estrada MP, Carpio Y. Novel IFNgamma homologue identified in Nile tilapia (Oreochromis niloticus) links with immune response in gills under different stimuli. Fish Shellfish Immunol. 2017 Dec;71:275-285. doi: 10.1016/j.fsi.2017.10.014. Epub 2017 Oct 7. PMID 29017941
- [Background] Aranake A, Mashour GA, Avidan MS. Minimum alveolar concentration: ongoing relevance and clinical utility. Anaesthesia. 2013 May;68(5):512-22. doi: 10.1111/anae.12168. Epub 2013 Feb 16. PMID 23414556
- [Background] Cho SY, Kwon YK, Nam M, Vaidya B, Kim SR, Lee S, Kwon J, Kim D, Hwang GS. Integrated profiling of global metabolomic and transcriptomic responses to viral hemorrhagic septicemia virus infection in olive flounder. Fish Shellfish Immunol. 2017 Dec;71:220-229. doi: 10.1016/j.fsi.2017.10.007. Epub 2017 Oct 7. PMID 29017947
- [Background] Tsilidis KK, Panagiotou OA, Sena ES, Aretouli E, Evangelou E, Howells DW, Al-Shahi Salman R, Macleod MR, Ioannidis JP. Evaluation of excess significance bias in animal studies of neurological diseases. PLoS Biol. 2013 Jul;11(7):e1001609. doi: 10.1371/journal.pbio.1001609. Epub 2013 Jul 16. PMID 23874156
- [Background] Zhu M, Tao Y, Pu J, Zhao H, Wan L, Zhang P, Tang C. Pharmacokinetics and Bioequivalence of Fudosteine in Healthy Chinese Volunteers Under Fasting and Fed Conditions: A 4-Way Replicate Crossover Study. Clin Pharmacol Drug Dev. 2023 Jan;12(1):30-37. doi: 10.1002/cpdd.1137. Epub 2022 Jul 6. PMID 35794358
- See also: the protocol of the study — http://pubmed.ncbi.nlm.nih.gov
- Available data/document: Study Protocol — http://www.chinadrugtrials.org.cn/clinicaltrials.searchlistdetail.dhtml — registered clinical trial about Brivaracetam oral solution on Chinese website